CLINICAL TRIAL: NCT00327028
Title: Randomised, Placebo Controlled, Double Blind, Parallel Group 3-Months Study of Phenytoin Efficacy in Bronchial Asthma Therapy
Brief Title: Study of Efficacy of Phenytoin in Therapy of Patients With Bronchial Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre of Chinese Medicine, Georgia (Other)
Collaborators: Rea Rehabilitation Centre, Georgia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTP-DP-0505-1205
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; Phenytoin, Diphenine; Antiepileptic drugs; Efficacy
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: Diphenine

SUMMARY:
The purpose of this study was evaluation the efficacy of antiepileptic drug phenytoin (diphenine) in the treatment of bronchial asthma.

DETAILED DESCRIPTION:
Effective therapy of asthma still remains quite serious problem. According current opinion of leading specialists, asthma is an inflammatory disorder. But asthma also is a paroxysmal disorder: many specialists underline paroxysmal clinical picture of asthma. According to some authors, neurogenic inflammation may play important role in asthma mechanism. But migraine and trigeminal neuralgia are also neurogenic inflammatory paroxysmal diseases, and some antiepileptic drugs, like diphenine and valproates, are very effective in therapy of these diseases - more than in 80% of cases. If bronchial asthma also is paroxysmal inflammatory disease, we can suppose a possibility that some antiepileptic drugs also may show high efficacy in asthma therapy. Taken in consideration this hypothesis, we performed a double-blind, placebo-controlled 3-month trial for evaluation of phenytoin (diphenine) efficacy in treatment of patients with bronchial asthma.

ELIGIBILITY:
Inclusion Criteria:

* Out patients
* Bronchial asthma has been known at least for 1 year
* Absence of long-term remissions of asthma (lasting more than 1 month)
* Poorly controlled asthma, due to various reasons
* Non-smokers

Exclusion Criteria:

* Presence of concomitant acute or chronic severe diseases
* Abnormal baseline haematology, blood chemistry or urinalysis
* Allergy or adverse reactions to investigational drug
* Age younger than 18 years old
* Long-term history of smoking
* Pregnancy or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61
Dates: Start 2005-09; Study Completion 2005-12

PRIMARY OUTCOMES:
At 3 months of treatment
Change from baseline of the PEFR and FEV1
Number of patients without asthma symptoms

SECONDARY OUTCOMES:
At 3 months of treatment
FEV1 before and after salbutamol inhalation
The daily (daytime and night-time) symptoms scores
Use of other antiasthmatic medication

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Tchelidze, MD, Study Director — CRO Evidence; Manana Pruidze, MD, PhD, Study Chair — Centre of Chinese Medicine; Merab Lomia, MD, PhD, Principal Investigator — "Rea" Rehabilitation Centre

REFERENCES:
- See also: Website of Neuroasthma Group — http://www.asthma.ge
- See also: Bronchial asthma as neurogenic paroxysmal inflammatory disease: a randomized trial with carbamazepine — http://www.ncbi.nlm.nih.gov/pubmed/16597501?ordinalpos=2&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum